CLINICAL TRIAL: NCT03320993
Title: Evaluación Del Impacto de la composición Nutricional de la Ingesta y Del Consumo de Alcohol en el Control glucémico Postprandial en Pacientes Con Diabetes Tipo 1
Brief Title: Impact of Meal Composition and Alcohol Consumption on Postprandial Glycemic Control in Subjects With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jorge Bondia (Other)
Collaborators: Hospital Francesc de Borja, Gandia, Spain (Unknown); Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Sponsor-Investigator, Jorge Bondia, Associate Professor, Universitat Politècnica de València
Organization: Universitat Politècnica de València (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: DPI2016-78831-C2-1-R_alcohol
Record Dates: First submitted 2017-10-20; First posted 2017-10-25 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: post-prandial glucose control; alcohol
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: 3-period, 3-treatment crossover design
Who Masked: Outcomes Assessor
Masking Description: Data analysis will be carried out by a person not involved in the study (she/he will be blind to the study condition)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Protein-Low Fat study (Active Comparator): Subjects will receive a mixed meal with carbohydrates (70g) plus a low content of proteins and fats
  Interventions: Other: Mixed meal with different macronutrient composition
- High Protein-High Fat study (Experimental): Subjects will receive a mixed meal with the same carbohydrates content of arm 1 (70g), but a greater amount of fats and proteins
  Interventions: Other: Mixed meal with different macronutrient composition
- High Protein-High Fat & alcohol study (Experimental): Subjects will receive the same mixed meal of the High Protein-High Fat study plus 0,7g of alcohol per Kg of weight
  Interventions: Other: Mixed meal with different macronutrient composition

INTERVENTIONS:
Other: Mixed meal with different macronutrient composition — A mixed meal with identical amount of carbohydrates but different content of protein, fat and alcohol will be given

SUMMARY:
Postprandial glucose control is a challenging issue in everyday diabetes care. Indeed, excessive postprandial glucose excursions are the major contributors to plasma glucose (PG) variability in subjects with type 1 diabetes (T1DM). In addition, the poor reproducibility of postprandial glucose response is burdensome for patients and healthcare professionals.

To date, the majority of prandial insulin dosing algorithms for subjects with T1DM considers only the carbohydrate (CHO) content of the meal. However, there is evidence (although with a certain degree of heterogeneity) that meal composition significantly affects postprandial glucose control, contributing to glycemic variability. Moreover, despite the high prevalence of alcohol consumption among patients with T1DM (about 30%, similar to that of the general population), data regarding its effect on the postprandial period are very limited.

This project will evaluate the effect of meal composition and alcohol consumption on postprandial glucose control in subjects with T1DM under intensive insulin treatment.

DETAILED DESCRIPTION:
Randomized, prospective, single-centre (Hospital Francesc de Borja, Gandia, Spain), single-blind (analysis), three -way, crossover study on type 1 diabetic subjects (n=12) under intensive insulin treatment.

Aim:

To assess the effect of mixed meal composition on postprandial glycemic control, in subjects with type 1 diabetes:

1. Combined effect of proteins and fats
2. Effect of alcohol consumption

Methods:

Each subject will undergo three mixed meal test studies (on three different days), with identical CHO content: On one occasion a low fat-low protein meal will be given, and on another a high fat-high protein one, both consumed with a non-alcoholic drink; on a third occasion the same high fat-high protein meal will be consumed, but this time accompanied by an equal volume of an alcoholic drink.

Patients will arrive at the research unit at 8:00 am and their blood glucose will be stabilized around 90 mg/dl before each mixed meal test. After the mixed meal, blood will be drawn every 5-30 min during a 6 hour post-prandial period to assess plasma glucose, hormones and metabolites concentration.

ELIGIBILITY:
Inclusion Criteria:

Patients with type 1 diabetes mellitus for more than one year, aged between 18 and 60 years; on intensive insulin therapy by means of CSII (continuous subcutaneous insulin infusion) or MDI (multiple daily injections) for at least 6 months before screening; glycosylated haemoglobin of 6-8.5%; without severe chronic micro- and macroangiopathic diabetic complications and with a body mass index (BMI) between 18 and 30 kg/m2.

Exclusion Criteria:

* Pregnancy and lactation
* Hypoglycemia unawareness
* Fatal or progressive disease
* Drugs or alcohol abuse
* HIV, active hepatitis B, active hepatitis C
* Hepatic disease (aminotransferases AST or ALT >2 times above normal)
* Clinically relevant microangiopathic disease, or other diseases that may interfere with participation in the study or data analysis
* Pre-planned surgery
* Blood donation in the previous 3 months for men and 6 months for women
* Mental conditions that may interfere with the subject's comprehension of the aims and possible consequences of the study
* Non-compliant subjects
* Use of experimental medications or devices during the previous 30 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Plasma Glucose | 6 hours (plasma glucose will be measured every 5-15 minutes during the 6-hour post-prandial period of each mixed meal test).
  Post-prandial plasma glucose time series

SECONDARY OUTCOMES:
AUC-PG | AUC of plasma glucose will be calculated for the whole 6 hour post-prandial period, for the early 0-3 hour post-prandial period and for the late 3-6 hour post-prandial period.
  Area Under the Curve (AUC) of Plasma Glucose in the 0-6h, 0-3h and 3-6h post-prandial periods

OTHER OUTCOMES:
Time in range | 6 hours (time in range during the 6 hour post-prandial period)
  Time in acceptable glucose range (70-180 mg/dl)
C Max | 6 hours (maximum plasma glucose concentration during the 6 hour post-prandial period)
  Maximum of plasma glucose concentration
T max | 6 hours (Time of maximum plasma glucose concentration during the 6 hour post-prandial period)
  Time of Maximum plasma glucose concentration
Hormones and metabolites | 6 hours (plasma hormones and metabolites will be measured every 30 minutes during the 6-hour post-prandial period)
  Plasma concentration of free fatty acids, beta-OH-butyrate, lactate, alanine, counterregulatory hormones

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Rossetti, PhD, Principal Investigator — Hospital Francesc de Borja, Gandia; Jorge Bondia Company, PhD, Study Director — Universitat Politècnica de València
Locations (1):
- Hospital Francesc de Borja, Gandia, Valencia, Spain

REFERENCES:
- [Background] Bell KJ, Smart CE, Steil GM, Brand-Miller JC, King B, Wolpert HA. Impact of fat, protein, and glycemic index on postprandial glucose control in type 1 diabetes: implications for intensive diabetes management in the continuous glucose monitoring era. Diabetes Care. 2015 Jun;38(6):1008-15. doi: 10.2337/dc15-0100. PMID 25998293
- [Background] Bell KJ, Toschi E, Steil GM, Wolpert HA. Optimized Mealtime Insulin Dosing for Fat and Protein in Type 1 Diabetes: Application of a Model-Based Approach to Derive Insulin Doses for Open-Loop Diabetes Management. Diabetes Care. 2016 Sep;39(9):1631-4. doi: 10.2337/dc15-2855. Epub 2016 Jul 7. PMID 27388474
- [Background] Barnard K, Sinclair JM, Lawton J, Young AJ, Holt RI. Alcohol-associated risks for young adults with Type 1 diabetes: a narrative review. Diabet Med. 2012 Apr;29(4):434-40. doi: 10.1111/j.1464-5491.2012.03579.x. PMID 22248115
- [Background] Turner BC, Jenkins E, Kerr D, Sherwin RS, Cavan DA. The effect of evening alcohol consumption on next-morning glucose control in type 1 diabetes. Diabetes Care. 2001 Nov;24(11):1888-93. doi: 10.2337/diacare.24.11.1888. PMID 11679452
- [Background] Kerr D, Cheyne E, Thomas P, Sherwin R. Influence of acute alcohol ingestion on the hormonal responses to modest hypoglycaemia in patients with Type 1 diabetes. Diabet Med. 2007 Mar;24(3):312-6. doi: 10.1111/j.1464-5491.2006.02054.x. PMID 17263767
- [Derived] Garcia A, Moscardo V, Ramos-Prol A, Diaz J, Boronat M, Bondia J, Rossetti P. Effect of meal composition and alcohol consumption on postprandial glucose concentration in subjects with type 1 diabetes: a randomized crossover trial. BMJ Open Diabetes Res Care. 2021 Oct;9(1):e002399. doi: 10.1136/bmjdrc-2021-002399. PMID 34620620